CLINICAL TRIAL: NCT00077350
Title: A Phase II Trial of Triapine® (NSC #663249) in Combination With Gemcitabine as Second Line Treatment of Non-Small Cell Lung Cancer
Brief Title: A Phase II Trial of Triapine (NSC #663249) in Combination With Gemcitabine as Second Line Treatment of Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02971; E1503; U10CA021115 (NIH); CDR0000350200 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; Gemcitabine

ARMS (1):
- Treatment (triapine and gemcitabine hydrochloride) (Experimental): Patients receive 3-AP (Triapine^®) IV over 2 hours and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: triapine; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as 3-AP and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving 3-AP together with gemcitabine may kill more tumor cells. This phase II trial is studying how well giving 3-AP together with gemcitabine works as second-line therapy in treating patients with progressive or recurrent non-small cell lung cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the antitumor response rate (by tumor measurement per the RECIST criteria) in patients taking this combination in the setting of second line treatment for NSCLC.

SECONDARY OBJECTIVES:

I. To evaluate the rate of stable disease, time to treatment progression, duration of response, and survival of patients taking this combination treatment.

II. To estimate the safety and tolerability of this combination in this phase II trial of patients with relapsed NSCLC.

TERTIARY OBJECTIVES:

I. To evaluate the potential effects of MDR polymorphisms in patients taking Triapine® in this combination.

II. To evaluate the effect of Triapine® and gemcitabine on RRM1, RRM2, and p53R2 protein expression per IHC and gene expression per RT-PCR from baseline diagnostic paraffin embedded blocks.

III. To evaluate both germline (peripheral blood) and tumor DNA for the presence of p53 mutations.

OUTLINE: This is a multicenter study.

Patients receive 3-AP (Triapine^®) IV over 2 hours and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for up to 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed non-small cell lung cancer (NSCLC); cytology alone is not acceptable
* Patients must have progressive or recurrent NSCLC, and must have failed one and only one prior cytotoxic chemotherapy regimen for advanced disease; patients must not have received prior gemcitabine chemotherapy
* Patients must have measurable disease, as defined by RECIST, within 4 weeks prior to registration
* Patients must have an ECOG performance status of 0 or 1
* Bilirubin < 1.5 x upper limit of normal
* AST (SGOT) < 3 x upper limit of normal
* Serum creatinine =< 1.5 mg/dL, or calculated creatinine clearance >= 60 mL/min
* Absolute granulocyte count >= 1500/mm3 and WBC >= 3000/mm^3
* Hemoglobin >= 9 g/L
* Platelet count >= 100,000/mm^3
* Patients must have completed any radiation therapy >= 3 weeks prior to registration
* Patients must have completed prior cytotoxic chemotherapy >= 3 weeks prior to registration and have recovered from adverse effects from the chemotherapy to =< Grade 1, or baseline
* Patients with brain metastases which have been treated are eligible if the patient is > 3 weeks post completion of treatment for their brain metastases, and patient is neurologically stable; patients with previous brain metastases who have not yet received therapy specifically intended for their brain metastases are not eligible to enroll in this protocol
* Life expectancy greater than 3 months
* Pregnant women are excluded from this study because Triapine® is a heterocyclic carboxaldehyde thiosemicarbazone with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Triapine®, breastfeeding should be discontinued if the mother is treated with Triapine®; women must not be pregnant or breastfeeding due to the absence of information regarding the use of these agents in these populations; a negative serum pregnancy test is required within 14 days of study entry; the effects of Triapine® on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because heterocyclic carboxaldehyde thiosemicarbazones as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination antiretroviral therapy are excluded from the study because of possible pharmacokinetic interactions with Triapine®
* Patients must not have an active second malignancy
* Patients must not have, at the time of registration, uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements; furthermore, since hypoxemia may cause serious adverse events in persons with serious cardiac and/or pulmonary disease, patients at the time of registration with a history of myocardial infarction within the prior 6 months, or with symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia requiring medical intervention (with the exception of chronic, stable, asymptomatic atrial fibrillation), or pulmonary disease requiring oxygen are excluded
* Patients must not have dementia or active psychosis
* Patients must not have used any investigational agent in the month before study enrollment
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Triapine® or other agents used in this study
* Patients must not have a clinical history of G6PD (glucose-6-phosphate dehydrogenase) deficiency; persons at high risk for this condition (patients of African, Asian, or Mediterranean origin/ancestry) must undergo specific clinical testing at protocol entry for this condition; patients testing positive for G6PD deficiency are excluded from protocol entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-07; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 1.5 years
  A true objective response rate of at least 25% will be considered evidence for further exploration of this regimen. A true response rate less than or equal to 5% will be considered evidence of minimal activity not worthy of further study.

SECONDARY OUTCOMES:
Rate of stable disease | Up to 1.5 years
Time to treatment progression | Up to 1.5 years
Duration of response | Up to 1.5 years
Overall survival | Up to 1.5 years
Toxicity using NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 | Up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anne Traynor, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States